CLINICAL TRIAL: NCT07146503
Title: ESKPSY: Esketamine in Real-World Settings: Clinical Outcomes, Predictors of Response, Life Functioning and Biological Pathways
Brief Title: Esketamine Nasal Spray in Real-World Settings in Treatment-Resistant Depression
Acronym: ESKPSY
Status: Recruiting | Type: Observational
Sponsor: Riccardo Guglielmo (Other)
Responsible Party: Sponsor-Investigator, Riccardo Guglielmo, Principal Investigator, Universita degli Studi di Genova
Organization: Universita degli Studi di Genova (Other)
Other Study IDs: D33C22001340002
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Depression and Quality of Life; Treatment Resistant Depression (TRD); Anhedonia; Apathy; Anxiety; Cognition; Temperament; Psychiatric Comorbidities
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant; Anhedonia; Lethargy; Anxiety Disorders | interventions — Esketamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Esketamine (Intranasal Spray) — Esketamine Intranasal Spray at a dosage ranging from 28 to 84 mg weekly, with twice-weekly administration during the first month of treatment, according to the approved labeling

SUMMARY:
This observational study investigates the use of Esketamine Intranasal Spray in patients with Treatment-Resistant Depression in Real-World Settings. The study aims to evaluate the clinical outcomes, including efficacy and safety, of esketamine treatment. It also explores predictors of treatment response, focusing on biological pathways such as genetics, neuroimaging, and psychophysical measures. Additionally, the study examines how esketamine impacts patients' life functioning, including social and occupational aspects. The goal is to better understand who benefits most from esketamine and how it affects daily life, to improve personalized care for patients with difficult-to-treat depression.

ELIGIBILITY:
Inclusion criteria were: (a) age 18-74, (b) DSM-5 diagnosis of a major depressive episode (MDE), (c) failure to respond to at least 2 prior antidepressant treatments (ADTs), and (d) current treatment with an SSRI or SNRI for which esketamine nasal spray was deemed appropriate.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Predictive Factors of Treatment Response: Biological, Clinical, and Social Dimensions | Time Frame: from enrollment to one year of treatment
  MADRS, HAM-D, HAM-A, TCI-R, BPRS, AES, SHAPS, EQ-5D-5L, BDI-II, WPAI-D, SDS, TEMPS

SECONDARY OUTCOMES:
Panel of genetic polymorphisms (SNPs) predictive of clinical response to esketamine in patients with treatment-resistant depression. | from enrollment to one year of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Briasco, MD, Principal Investigator — Unige; Elisa Cavanna, MD, Principal Investigator — Unige; Riccardo Guglielmo, MD, Study Chair — Unige; Gianluca Serafini, MD, Study Director — Unige
Locations (4):
- Italy (4):
  - Ospedale Policlinico San Martino, Genova, Ge
  - Csm Dds 8, Genova, Ge
  - Università di Chieti, Chieti
  - ASST Fatebenefratelli Sacco, Milan

REFERENCES:
- [Result] Guglielmo R, Marino M, Briasco E, Cavanna E, Inuggi A, Schiavon F, Giacomini G, Malagamba D, Escelsior A, Martinotti G, Amore M, Serafini G. Predictors of Esketamine Response in Treatment-Resistant Depression: The Role of Temperament and Cumulative Treatment Resistance. CNS Drugs. 2025 Nov;39(11):1187-1191. doi: 10.1007/s40263-025-01210-7. Epub 2025 Aug 2. No abstract available. PMID 40751860

DOCUMENTS (1):
  • Study Protocol (2025-08-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT07146503/Prot_000.pdf